CLINICAL TRIAL: NCT02583919
Title: Double Blind, Randomized, Placebo-Controlled, Phase 2 Study to Evaluate the Safety, Tolerability and Efficacy of ISIS 449884 Administered Once Weekly for 26 Weeks in Patients With Type 2 Diabetes Being Treated With Metformin
Brief Title: Safety, Tolerability and Efficacy of ISIS-GCGRRx in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 449884-CS4
Record Dates: First submitted 2015-10-12; First posted 2015-10-22 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ISIS-GCGRRx - Dose Level 1 (Experimental): ISIS-GCGRRx - Dose Level 1
  Interventions: Drug: ISIS-GCGRRx- Dose Level 1
- ISIS-GCGRRx - Dose Level 2 (Experimental): ISIS-GCGRRx - Dose Level 2
  Interventions: Drug: ISIS-GCGRRx- Dose Level 2
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISIS-GCGRRx- Dose Level 1 — once weekly dosing for 26 weeks
  Other Names: Isis 449884
  Arms: ISIS-GCGRRx - Dose Level 1
Drug: ISIS-GCGRRx- Dose Level 2 — once weekly dosing for 26 weeks
  Other Names: Isis 449884
  Arms: ISIS-GCGRRx - Dose Level 2
Drug: Placebo — once weekly dosing for 26 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of ISIS-GCGRRx in combination with metformin versus placebo

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 75
* BMI ≥ 25.0 kg/m2
* HbA1c ≥ 8.0% and ≤ 10.5%
* Type 2 Diabetes Mellitus and on stable dose of Metformin
* Agree to conduct home-based (fasted) blood glucose testing as directed

Exclusion Criteria:

* Clinically significant abnormalities in medical history of physical exam
* Show evidence of uncorrected hypothyroidism or hyperthyroidism hormone results
* History of solid organ transplant or renal dialysis
* History of liver disease
* History of greater than 3 episodes of severe hypoglycemia within 6 months of screening
* Treatment with any other antidiabetic drug(s) other than metformin within 3 months of screening
* History of diabetic ketoacidosis
* Any other significant illness or condition that may interfere with the patient participating or completing the study
* Inability or unwillingness to comply with protocol or study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C | Week 27 and subsequent timepoints
  Change from Baseline

SECONDARY OUTCOMES:
Safety and Tolerability will be assessed by determining the incidence, severity, dose-relationship adverse-effects, and changes in laboratory evaluations within each dose cohort | 50 weeks
  Safety results in patients dosed with Isis 449884 will be compared with those from patients dosed with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Bhanot, Study Director — Ionis Pharmaceuticals, Inc.
Locations (17):
- United States (17):
  - Ionis Investigational Site, Greenbrae, California
  - Ionis Investigational Site, Huntington Park, California
  - Ionis Investigational Site, La Mesa, California
  - Ionis Investigational Site, Los Angeles, California
  - Isis Investigational Site, Spring Valley, California
  - Ionis Investigational Site, Port Orange, Florida
  - Ionis Investigational Site, Marietta, Georgia
  - Ionis Investigational Site, Oxon Hill, Maryland
  - Ionis Investigational Site, New York, New York
  - Ionis Investigational Site, Greensboro, North Carolina
  - Ionis Investigational Site, Morehead City, North Carolina
  - Ionis Investigational Site, Cincinnati, Ohio
  - Ionis Investigational Site, Eugene, Oregon
  - Ionis Investigational Site, Spartanburg, South Carolina
  - Ionis Investigational Site, Houston, Texas
  - Ionis Investigational Site, Katy, Texas
  - Ionis Investigational Site, Olympia, Washington

REFERENCES:
- [Derived] Morgan ES, Tai LJ, Pham NC, Overman JK, Watts LM, Smith A, Jung SW, Gajdosik M, Krssak M, Krebs M, Geary RS, Baker BF, Bhanot S. Antisense Inhibition of Glucagon Receptor by IONIS-GCGRRx Improves Type 2 Diabetes Without Increase in Hepatic Glycogen Content in Patients With Type 2 Diabetes on Stable Metformin Therapy. Diabetes Care. 2019 Apr;42(4):585-593. doi: 10.2337/dc18-1343. Epub 2019 Feb 14. PMID 30765435